CLINICAL TRIAL: NCT03965455
Title: Clinical Efficacy of Conventional and Diode Laser-Assisted Frenectomy in Patients With Abnormal Different Frenum Insertions: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-164
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Frenulum; Elongation
Keywords: labial frenum; laser therapy; recurrence; oral hyigiene
MeSH Terms: conditions — Recurrence | interventions — Lasers, Semiconductor; Oral Frenectomy; Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- conventional group
  Interventions: Procedure: Conventional
- diode laser group
  Interventions: Device: Diode laser

INTERVENTIONS:
Device: Diode laser — In the laser-assisted frenectomy, a diode laser device (GIGA Cheese II®, China) (λ= 810 nm) with a 400 µm diameter, plain-ended optical ﬁber tip was used for the procedure maintaining contact with oral mucosa at 2,5 W, 70 Hz frequency with a short pulse (140 microseconds) duration.
  Other Names: frenectomy
  Groups: diode laser group
Procedure: Conventional — In the conventional frenectomy, the incisions were applied using a scalpel blade no.15 on the upper and lower surface of the haemostat until the frenum was excised.
  Other Names: frenectomy
  Groups: conventional group

SUMMARY:
Aim: The aim of this retrospective study was to assess the frenum attachment recurrence and evaluate clinical parameters after conventional and diode laser-assisted frenectomy in patients with different abnormal frenum insertions.

Methods: Data records of 429 patients treated with maxillary labial frenectomy between January 1, 2016 and January 1, 2018 were screened. Records of 70 patients meeting the inclusion criteria were evaluated. Data were analyzed in terms of gender, age, category of frenum, presence of diastema, operation technique, type of periodontal disease. The distance between frenum attachment and mucogingival junction (FMGJ), plaque index (PI), gingival index (GI) and probing depth were assessed.

ELIGIBILITY:
Inclusion Criteria:

(a) systemically healthy, (b) nonsmoker, (c) aged between 18 and 65 years, (d) received initial periodontal treatment before frenectomy, (e) presence of central and lateral incisors and canines at maxilla, (f) not received any kind of periodontal surgery, prosthodontic and restorative treatment which may affect the anatomy of the relevant region.

Exclusion Criteria:

Subjects with incomplete documentation and without at least 6-week follow-up observation were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study utilized treatment records of patients treated with maxillary labial frenectomy in the Clinics of Periodontology, Faculty of Dentistry, Marmara University.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
recurrence | 6 weeks
  Recurrence is evaluated by the formation of an intact mucosa with the frenum attached to its new position

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)